CLINICAL TRIAL: NCT03426150
Title: In Situ Effect of Casein Phosphopeptide--amorphous Calcium Phosphate on the Surface Microhardness of Human Enamel Subjected to in Vivo Acid Attacks
Brief Title: Casein Phosphopeptide--amorphous Calcium Phosphate on Human Enamel Subjected to in Vivo Acid Attacks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Hao Yu, Department Head, Fujian Medical University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 20151225
Record Dates: First submitted 2018-01-24; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Dental Erosion
MeSH Terms: conditions — Tooth Erosion | interventions — casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPP-ACP (Experimental): Tooth mousse (GC, Japan) application on the specimen surface for 3 min.
  Interventions: Drug: CPP-ACP
- Deionized water (Placebo Comparator): Deionized water application on the specimen surface for 3 min
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: CPP-ACP — The surfaces of specimens were pretreated with CPP-ACP for 3 min
  Arms: CPP-ACP
Drug: Placebos — The surfaces of specimens were pretreated with deionized water for 3 min
  Arms: Deionized water

SUMMARY:
40 specimens were prepared from fresh-extracted human molars and further embedded using the acrylic resin. Specimens were randomly divided into 2 groups according to the treatment before in vivo erosion (n=20): CPP-ACP for 3 min (CPP-ACP group) and deionized water for 3 min (control group). 10 healthy volunteers were recruited and customized maxillary appliance containing 4 specimens (2 from CPP-ACP group and 2 from control group) was fabricated for each volunteer. Participants were instructed to drink 150 ml cola in 5 min using the gargling method after placing appliances intraorally for 2 h. The in vivo attacks were performed 4 X 5 min with 1-h interval daily over 7 d. The surface microhardness and surface microstructure of the specimens were evaluated at the baseline and after the treatment. The data were statistically analyzed using three-way ANOVA and post hoc tests. Data were considered statistically significant at a level of P <0.05.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years of age and in good general health
* Dental erosion and wear degree is 0-1

Exclusion Criteria:

* Systemic diseases or oral mucosal disorders
* Current orthodontic treatment
* Pregnancy
* Known allergies to the experimental drink
* Had been given drugs which lead to dry oral more regularly within half a year

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-12-25 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
Surface microhardness | baseline
  a Vickers microhardness tester with microscopic lens was used, with a 100 g load and 30-s dwell time. Three microhardness measurements were obtained on the top surface of each specimen.
Surface microhardness | 7 days
  a Vickers microhardness tester with microscopic lens was used, with a 100 g load and 30-s dwell time. Three microhardness measurements were obtained on the top surface of each specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Yu, DDS, PhD, Principal Investigator — School and Hospital of Stomatology, Fujian Medical University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yu H, Jiang NW, Ye XY, Zheng HY, Attin T, Cheng H. In situ effect of Tooth Mousse containing CPP-ACP on human enamel subjected to in vivo acid attacks. J Dent. 2018 Sep;76:40-45. doi: 10.1016/j.jdent.2018.05.021. Epub 2018 May 30. PMID 29857075